CLINICAL TRIAL: NCT06927219
Title: Web-Based Data Collection Through the Research Accelerated by You (RAY) Lupus Registry
Brief Title: Research Accelerated by You Lupus Registry
Acronym: RAY
Status: Recruiting | Type: Observational
Sponsor: Lupus Foundation of America (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00020515
Record Dates: First submitted 2025-03-12; First posted 2025-04-15 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus (SLE); Lupus Nephritis (LN); Cutaneous Lupus Erythematosus (CLE)
Keywords: lupus; registry
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis; Lupus Erythematosus, Cutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lupus Patients: This is an observational study of people living with systemic lupus erythematosus, lupus nephritis, cutaneous lupus erythematosus or a mixture of these diseases

SUMMARY:
Summary The Lupus Foundation of America (LFA) Research Accelerated by You (RAY) Registry is a fully remote, longitudinal registry designed to collect data from adults and children living with lupus. The primary goal is to better understand the diagnosis, treatment, care, and quality of life for those affected by the disease.

Remote Participation This is a decentralized, online-only registry. Participation is conducted entirely through a secure web-based portal. There are no physical site visits or travel requirements; participants can contribute from any location with internet access.

Participation Details

Consent: Informed consent is completed electronically.

Surveys: Participants complete electronic surveys upon enrollment and every six months thereafter.

Data Types: Collected data is self-reported and includes demographics, diagnosis history, treatment information, and patient-reported outcomes (PROs), such as quality of life.

Purpose and Data Use The LFA uses registry data to:

Address Constituent Needs: Inform programs and resources for the lupus community.

Advance Research: Share patient insights with to ensure therapies are developed with the consideration of what matters and what matters most to people living with lupus.

Patient Engagement and Clinical Research Matching: Participants may be contacted to assess eligibility for patient engagement or clinical research opportunities or to complete specific sub-surveys regarding trial participation.

DETAILED DESCRIPTION:
This is a multinational, direct-to-patient registry available to patients in the United States and Canada. The registry will enroll 10,000 people living with lupus who have a diagnosis of:

* Systemic Lupus Erythematosus
* Lupus Nephritis (Lupus Related Kidney Disease)
* Skin-Only Lupus (Cutaneous Lupus)
* Skin-Only Lupus With Scarring (Discoid Lupus)
* Lupus Caused By Medication(S) (Drug-Induced Lupus)

The registry will include questions about demographics, diagnostic journey, signs and symptoms, treatments, impact of lupus on health and quality of life, patient report outcomes and preferences related to clinical trials. The registry will also collect information about fatigue and work productivity.

ELIGIBILITY:
Inclusion Criteria:

* For adults with lupus, the individual who completes the Registry:

  * is 18 years of age or older
  * has a self-reported diagnosis of lupus by a physician or health care provider
  * is willing and able to provide informed consent
  * is able to read and understand English sufficiently to complete the survey questions
  * has access to a computer with an internet connection

For children under 18 with lupus, the individual who completes the Registry is:

* 18 years of age or older
* the parent/legal guardian/legally authorized representative of a child under 18 years of age that has a diagnosis of lupus by a physician or health care provider
* willing and able to provide consent for the child under 18 years of age and to obtain assent from the child between 7-17 years of age
* able to access a computer with an internet connection
* able to read and understand English sufficiently to complete the survey questions

For adults with lupus unable to provide consent, the individual who completes the Registry is:

* 18 years of age or older
* the legally authorized representative of an adult 18 or older who is unable to provide consent and has a diagnosis of lupus by a physician or health care provider
* willing and able to provide consent for the adult with lupus
* able to access a computer with an internet connection
* able to read and understand English sufficiently to complete the survey questions

Exclusion Criteria:

* People who are not living with lupus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People diagnosed with systemic lupus erythematosus, lupus nephritis (lupus-related kidney disease), Cutaneous lupus erythematosus (CLE) or discoid lupus erythematosus (DLE)
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Chronic Illness Therapy-Fatigue Scale | Over a 10 year period
  This 13-item scale measures self-report fatigue and impacts on activities of daily living and functioning. The scale as been validated in various disease areas including cancer patients, cancer survivors, rheumatoid arthritis and systemic lupus erythematosus.
Work Productivity and Activity Impairment | Over a 10 year period.
  This outcome measure evaluates impairments over the past 7 days in both paid and unpaid work due to an individual's health.

CONTACTS AND LOCATIONS:
Overall Officials: Joy N Buie, PhD, MSCR, RN, Principal Investigator — Lupus Foundation of America
Locations (1):
- Online Registry - No Physical Site Required, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No